CLINICAL TRIAL: NCT00535795
Title: A Phase III Study to Assess Conventional RT w/ Conventional Plus Accelerated Boost RT in the Treatment of Nasopharyngeal CA
Brief Title: Phase III: Assess Conventional RT w/ Conventional Plus Accelerated Boost RT in the Treatment of Nasopharyngeal CA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAC#0971-004
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2011-12

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Conventional Radiation Therapy (XRT), one fraction per day, from Sunday to Thursday every week.
  Interventions: Radiation: Radiation Therapy
- 2 (Experimental): Conventional Plus accelerated boost Radiation Therapy (XRT), from Sunday to Thursday every week.
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — Radiation Therapy

SUMMARY:
Phase III: Assess conventional RT w/ conventional Plus accelerated boost RT in the treatment of nasopharyngeal CA

DETAILED DESCRIPTION:
It's a phase III study to assess conventional Rad Therapy with conventional Plus accelerated boost Rad Therapy in the treatment of nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with nasopharyngeal Carcinoma

Exclusion Criteria:

* Patients with carcinoma other than histo-pathologically confirmed nasopharyngeal CA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
safety and efficacy | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Nasser Al Rajhi, MD, Principal Investigator — KFSH&RC
Locations (1):
- KFSH&RC, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided